CLINICAL TRIAL: NCT04881487
Title: A Randomized Controlled Trial on Additional Treatment for Isolated Local Pancreatic Cancer Recurrence Using Stereotactic Body Radiation Therapy
Brief Title: Additional Treatment for Isolated Local Pancreatic Cancer Recurrence Using Stereotactic Body Radiation Therapy
Acronym: ARCADE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Pancreatic Cancer Group (DPCG) (Unknown)
Responsible Party: Principal Investigator, Martijn P.W. Intven, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL74336.041.20; 20-805 (Other: METC Utrecht); 12568 (Other Grant/Funding Number: KWF)
Record Dates: First submitted 2021-03-25; First posted 2021-05-11 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Pancreatic Ductal Adenocarcinoma
Keywords: Stereotactic body radiation therapy

STUDY DESIGN:
Intervention Model Description: Trials within Cohorts (TwiCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional stereotactic body radiation therapy (Experimental): SBRT in addition to standard of care.
  Interventions: Radiation: Additional stereotactic body radiation therapy
- Standard of care (No Intervention): Treatment according to current clinical practice.

INTERVENTIONS:
Radiation: Additional stereotactic body radiation therapy — 5 fractions of 8 Gray stereotactic body radiation therapy in addition to standard of care.
  Arms: Additional stereotactic body radiation therapy

SUMMARY:
A randomized controlled trial, nested within an existing prospective cohort (Dutch Pancreatic Cancer Project; PACAP) according to the 'trials within cohorts' (TwiCs) design in which the effect of additional local ablative therapy compared to current standard of care alone, on survival after recurrence in patients with isolated local pancreatic ductal adenocarcinoma (PDAC) recurrence. The most important secondary endpoint is quality of life. Other secondary endpoints are treatment response, acute and late toxicity, overall survival, progression-free survival, local progression-free survival, distant metastases free survival and reasons for non-eligibility or exclusion.

DETAILED DESCRIPTION:
Rationale: Disease recurrence remains the main cause of mortality in patients who underwent resection for PDAC. In case of recurrence, patients are currently treated with palliative chemotherapy or best supportive care. In 20-30% of all patients, isolated local PDAC recurrence occurs after resection, which is frequently associated with considerable morbidity from local destructive tumor growth. Although survival after recurrence is predominantly determined by systemic disease, additional local ablative therapy might be of value to improve local disease control in these patients, which could positively affect survival and quality of life (QoL). Previously, radiation therapy has played only a minor role in the treatment of PDAC. As the pancreas is tightly surrounded by organs with limited radiation dose tolerance and subjected to abdominal motion due to respiration and peristalsis, optimal dose delivery has been impeded with conventional radiotherapy techniques. The development of image-guided stereotactic body radiation therapy (SBRT) techniques, however, enabled safe delivery of high irradiation doses to pancreatic lesions. Early retrospective studies have suggested that SBRT might lead to improved local control in patients with isolated local PDAC recurrence, potentially having a beneficial effect on both survival and QoL. In the current, multicenter randomized controlled trial, the value of SBRT in addition to standard of care in patients with isolated local PDAC recurrence is compared to standard of care alone, with regard to both survival and quality of life outcomes.

Objective: The main objective of this study is to improve survival after recurrence in patients with isolated local PDAC recurrence using local ablative treatment with SBRT in addition to standard of care. Furthermore, the effects of additional SBRT on QoL will be evaluated within this study.

Study design: A randomized controlled trial, nested within a prospective cohort (PACAP) according to the TwiCs design.

Study population: PACAP-participants with isolated local PDAC recurrence after primary resection who provided informed consent for being randomized in future studies.

Intervention: Local ablative therapy (5 times 8 Gray SBRT) in addition to standard of care.

Comparison: standard of care.

Main study endpoints: The main study endpoint is survival after recurrence. The most important secondary endpoint is quality of life. Other secondary endpoints are radiological treatment response, acute and late toxicity, overall, progression-free, local progression-free and distant metastasis free survival and reasons for non-eligibility or exclusion.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the PACAP cohort with written informed consent for being randomized in future studies
* Isolated local recurrence after primary PDAC resection
* Minimum age of 18 years

Exclusion Criteria:

* Distant metastases
* Expected lifespan < 3 months
* Ineligibility for MRI or CT according to the protocol of the local radiology department;
* Highly selective cases with resectable, isolated local recurrence without the need for either systemic or local ablative induction therapy, eligible for re-resection according to the expert panel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Survival after recurrence | From the date of PDAC recurrence diagnosis until either death from any cause or last follow-u, whichever came first, assessed up to 24 months
  The interval between the date of PDAC recurrence diagnosis and either death from any cause or last follow-up.

SECONDARY OUTCOMES:
Patient reported Quality of Life as assessed using Exocrine Pancreatic Insufficiency (EPI) questionnaire | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP-cohort. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP-participants.
Patient reported non-disease specific health-related Quality of Life (HRQoL) as assessed using the EQ-5D-5L | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP-cohort. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP-participants.
Patient reported cancer-specific HRQoL as assessed using the EORTC QLQ-C30 | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP-cohort. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP-participants.
Patient reported tumor-specific HRQoL as assessed using the EORTC LQPAN26 | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP-cohort. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP-participants.
Patient reported chemotherapy-induced peripheral neuropathy as assessed using the EORTC QLQ-CIPN20 | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP-cohort. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP-participants.
Patient reported Quality of Life as assessed using the happiness, hospital, anxiety and depression scale (HADS) | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP-cohort. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP-participants.
Patient reported Quality of Life as assessed using the worry of progression of cancer scale (WOPS) | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP-cohort. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP-participants.
Treatment response assessed on CT-imaging (graded according to RECIST guidelines) | During and immediately after the intervention (SBRT treatment)
  Response to SBRT treatment.
Acute and late toxicity of SBRT as assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Through study completion, an average of 18 months
  Assessed during regular follow-up moments. In the intervention arm acute toxicity will be monitored by the treating radiation oncologist. Acute toxicity will be defined as toxicity within 90 days from the end of SBRT treatment and will be assessed in week 1, 3, 6 and 12. Late toxicity is defined as toxicity occurring > 90 days from SBRT.
Overall survival | From the date of primary resection until the date of death from any cause or last follow-up, whichever came first, assessed up to 18 months
  The interval between the date of primary resection and the date of death from any cause or last follow-up.
Progression-free survival | From the date of disease recurrence until the date that local and/or distant progression of disease occurs, assessed up to 18 months
  The interval between the date of disease recurrence and the date that local and/or distant progression of disease occurs.
Local progression-free survival | From the date of disease recurrence until the date that locoregional progression of disease occurs, assessed up to 18 months
  The interval between the date of disease recurrence and the date that locoregional progression of disease occurs.
Distant metastases free survival | From the date of disease recurrence until the date that distant progression of disease occurs, assessed up to 18 months
  The interval between the date of disease recurrence and the date that distant progression of disease occurs.
Reasons for non-eligibility or exclusion for SBRT treatment | At the time the patient is assessed eligible for the intervention. Assessed through the study, up to 18 months
  e.g. poor condition, patients wish, deteriorated condition, age.

CONTACTS AND LOCATIONS:
Overall Officials: M. P.W. Intven, MD, PhD, Principal Investigator — Regional Academic Cancer Center Utrecht (RACU); A. M.E. Bruynzeel, MD, PhD, Principal Investigator — Amsterdam University Medical Center, VUmc; J. Nuyttens, MD, PhD, Principal Investigator — Erasmus Medical Center; I. Q. Molenaar, MD, PhD, Principal Investigator — Regional Academic Cancer Center Utrecht (RACU); M. G.H. Besselink, MD, PhD, Principal Investigator — Amsterdam University Medical Center, AMC; B. Groot Koerkamp, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - Amsterdam University Medical Center, VUmc, Amsterdam, North Holland
  - Erasmus University Medical Center, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
De-identified data generated during the ARCADE trial will be made available to other researcher upon request from M.P.W. Intven.
Supporting Information: Study Protocol
Access Criteria: Upon request.

REFERENCES:
- [Derived] van Goor IWJM, Daamen LA, Besselink MG, Bruynzeel AME, Busch OR, Cirkel GA, Groot Koerkamp B, Haj Mohammed N, Heerkens HD, van Laarhoven HWM, Meijer GJ, Nuyttens J, van Santvoort HC, van Tienhoven G, Verkooijen HM, Wilmink JW, Molenaar IQ, Intven MPW; Dutch Pancreatic Cancer Group. A nationwide randomized controlled trial on additional treatment for isolated local pancreatic cancer recurrence using stereotactic body radiation therapy (ARCADE). Trials. 2022 Oct 28;23(1):913. doi: 10.1186/s13063-022-06829-1. PMID 36307892